CLINICAL TRIAL: NCT00005039
Title: A Phase II Randomized Trial of Recombinant Fowlpox and Recombinant Vaccinia Virus Expressing PSA in Patients With Adenocarcinoma of the Prostate
Brief Title: Vaccine Therapy in Treating Patients With Advanced Adenocarcinoma of the Prostate (Prostate Cancer)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02319; DFHCC 98-262; U01CA062490 (NIH); CDR0000067630 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PROSTVAC

ARMS (2):
- Arm I (Experimental): Patients receive recombinant fowlpox-PSA vaccine IM at the MTD from the safety cohort every 4 weeks for 3 courses. Patients then receive recombinant vaccinia-PSA vaccine intradermally every 4 weeks for 2 courses.
  Interventions: Biological: recombinant fowlpox-prostate specific antigen vaccine; Biological: recombinant vaccinia prostate-specific antigen vaccine; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients receive the same vaccines as in arm I but in reverse order.
  Interventions: Biological: recombinant fowlpox-prostate specific antigen vaccine; Biological: recombinant vaccinia prostate-specific antigen vaccine; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: recombinant fowlpox-prostate specific antigen vaccine — Given IM
  Other Names: fowlpox-PSA vaccine; recombinant fowlpox-PSA vaccine; rF-PSA
Biological: recombinant vaccinia prostate-specific antigen vaccine — Given intradermally
  Other Names: Prostate Specific Antigen Expressing Vaccinia Virus Vaccine; rV-PSA vaccine; vaccinia prostate-specific antigen vaccine; vaccinia-prostate-specific antigen vaccine; VPSA
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Randomized phase II trial to determine the effectiveness of vaccine therapy in treating patients who have advanced adenocarcinoma of the prostate (prostate cancer). Vaccines made from a person's prostate cancer cells may make the body build an immune response to kill tumor cells

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the toxicity and maximum tolerated dose of recombinant fowlpox prostate-specific antigen (PSA) vaccine in patients with advanced adenocarcinoma of the prostate.

II. Determine whether vaccination with recombinant fowlpox-PSA vaccine is associated with antitumor activity in these patients.

III. Determine the efficacy of prime and boost regimens using recombinant fowlpox-PSA vaccine and recombinant vaccinia-PSA vaccine in these patients.

IV. Compare the PSA-specific T-cell response in patients treated with recombinant fowlpox-PSA vaccine followed by recombinant vaccinia-PSA vaccine vs the same vaccines but in reverse order.

OUTLINE: This is a randomized, open-label, multicenter, dose-escalation study of recombinant fowlpox prostate-specific antigen (PSA) vaccine.

SAFETY COHORT: The first cohort of 3 patients receives vaccination with recombinant fowlpox-PSA vaccine intramuscularly (IM). Treatment repeats every 4 weeks for 3 courses. In the absence of unacceptable toxicity in the first cohort, the second cohort of 3 patients receives the same vaccine at the dose level immediately higher than the first cohort dose level. In the presence of unacceptable toxicity in the first cohort, the second cohort of 3 patients receives the same vaccine at a dose level lower than the first cohort dose level. The maximum tolerated dose (MTD) is the dose preceding that at which 1 of 6 patients experiences grade 3 or worse dose-limiting toxicity.

Subsequent patients are assigned to one of two vaccination groups based on prior treatment with recombinant vaccinia-PSA vaccine:

GROUP A (no prior recombinant vaccinia-PSA vaccine): Patients are randomized to one of two vaccination arms:

ARM I: Patients receive recombinant fowlpox-PSA vaccine IM at the MTD from the safety cohort every 4 weeks for 3 courses. Patients then receive recombinant vaccinia-PSA vaccine intradermally every 4 weeks for 2 courses.

ARM II: Patients receive the same vaccines as in arm I but in reverse order.

GROUP B (prior recombinant vaccinia-PSA vaccine): Patients receive treatment as in arm I, group A.

GROUPS A AND B: Patients with stable or responding disease at 6 months after completion of vaccination therapy may continue treatment on the group and arm to which they were originally assigned. Treatment repeats every 6-9 months in the absence of disease progression.

Patients are followed monthly for 6 months and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate with evidence of metastatic disease including any of the following:

  * Lymph node positive and prostate-specific antigen (PSA) at least 10 ng/mL
  * Bone scan positive and PSA at least 10 ng/mL
  * Prior radical prostatectomy with rising PSA and PSA at least 2 ng/mL
  * Prior radiotherapy and PSA at least 10 ng/mL
  * Prior cryosurgery and PSA at least 10 ng/mL

    * PSA criteria does not apply to patients who are assigned to group B of this study and were previously treated on vaccine trial DFCI-96079
* No symptomatic metastatic disease (no bony pain)
* Complete HLA typing required
* Performance status - ECOG 0 or 1
* WBC greater than 2,000/mm^3
* Platelet count greater than 100,000/mm^3
* Bilirubin less than 2.0 mg/dL
* SGPT less than 4 times upper limit of normal
* Creatinine less than 4.0 mg/dL
* No altered immune function such as eczema
* No autoimmune diseases such as the following:

  * Autoimmune neutropenia, thrombocytopenia, or hemolytic anemia
  * Systemic lupus erythematosus, Sjögren's syndrome, or scleroderma
  * Myasthenia gravis
  * Goodpasture's syndrome
  * Addison's disease, Hashimoto's thyroiditis, or active Graves' disease
* HIV negative
* No allergy or untoward reaction to prior vaccinia (smallpox) vaccination
* No hypersensitivity to eggs
* No prior or concurrent extensive eczema or skin disorders (e.g., extensive psoriasis, burns, impetigo, or disseminated zoster)
* No other concurrent serious illness
* No active infection requiring antibiotics until infection has cleared and antibiotics have been stopped for at least 3 days
* Fertile patients must use effective contraception
* No close contact or household contact with the following high-risk individuals for at least 2 weeks after each vaccination:

  * Children under age 5
  * Pregnant or nursing women
  * Individuals with prior or concurrent extensive eczema or other eczematoid skin disorders
  * Individuals with other acute, chronic, or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds)
  * Immunodeficient or immunosuppressed individuals (by disease or therapy) such as those with HIV infection
* See Disease Characteristics
* See Endocrine therapy
* Prior vaccinia (smallpox) immunization required
* No other concurrent biologic therapy (e.g., interferon or interleukin) for cancer
* No prior chemotherapy for metastatic disease
* No concurrent anticancer chemotherapy
* No prior hormonal therapy for metastatic disease
* Prior neoadjuvant hormonal therapy followed by prostatectomy or radiotherapy allowed
* Patients previously treated with recombinant vaccinia-PSA vaccine may have hormonal therapy since discontinuing that treatment (Group B)
* No concurrent hormonal therapy or steroids
* See Disease Characteristics
* See Endocrine therapy
* No concurrent radiotherapy
* See Disease Characteristics
* See Endocrine therapy
* No prior splenectomy
* At least 3 days since prior antibiotics
* No concurrent immunosuppressive treatment (e.g., after organ transplantation)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2000-01; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
PSA response | Up to 3 months after the final vaccine dose
  PSA response is assessed at 3 successive monthly determinations, starting 28 days after the final vaccine dose.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Paul Eder, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States